CLINICAL TRIAL: NCT02342392
Title: Intralesional Ranibizumab on Pterygium Vascularity, Size and Recurrence Rate: a Pilot Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Hao Chi Ho, DR., Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Pterygium
Keywords: pterygium; ranibizumab; anti-VEGF; recurrence; vascularity; size
MeSH Terms: conditions — Pterygium; Recurrence | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment group (Active Comparator): intralesional ranibizumab injected
  Interventions: Drug: ranibizumab
- control group (No Intervention): no intralesional ranibizumab injected.

INTERVENTIONS:
Drug: ranibizumab — Intralesional ranibizumab 0.3 mg/0.03mL injected 1 week before pterygium excision surgery.
  Other Names: Lucentis
  Arms: treatment group

SUMMARY:
The purpose of this study is to evaluate the pterygium vascularity and size before and after intralesional ranibizumab injection and to evaluate its recurrence rate following pterygium excision surgery.

DETAILED DESCRIPTION:
The purpose of this study is to:

1. Compare the vascularity of primary pterygium before and 1 week after intralesional ranibizumab (0.3 mg/0.03 mL) injection.
2. Compare the size of primary pterygium before and 1 week after intralesional ranibizumab (0.3 mg/0.03 mL) injection.
3. Compare the recurrence rate at 1 year after pterygium excision surgery between the group with and without intralesional ranibizumab injection.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary pterygium.
* Grade T3 (fleshy) pterygium.

Exclusion Criteria:

* Patients with other ocular surface disorders.
* Previous ocular surgery or trauma.
* History of systemic thromboembolic event.
* Pregnant women and lactating mother.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
pterygium recurrence | 1 year
  pterygium recurrence is defined as true recurrence with a fibrovascular tissue invading the cornea (grade 4 lesion)

SECONDARY OUTCOMES:
pterygium vessel area | 1 week
  Pterygium vesel area is defined as the as the ration of pixels occupied by the vessels within the pterygium area in percentage.
corneal pterygium area | 1 week
  Corneal pterygium area is defined as the as the ration of pixels occupied by the pterygium within the cornea area in percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chi Ho, MD, Principal Investigator — Hospital Universiti Sains Malaysia

REFERENCES:
- [Background] Lee DH, Cho HJ, Kim JT, Choi JS, Joo CK. Expression of vascular endothelial growth factor and inducible nitric oxide synthase in pterygia. Cornea. 2001 Oct;20(7):738-42. doi: 10.1097/00003226-200110000-00013. PMID 11588427
- [Background] Blaudschun R, Sunderkotter C, Brenneisen P, Hinrichs R, Peters T, Schneider L, Razi-Wolf Z, Hunzelmann N, Scharffetter-Kochanek K. Vascular endothelial growth factor causally contributes to the angiogenic response upon ultraviolet B irradiation in vivo. Br J Dermatol. 2002 Apr;146(4):581-7. doi: 10.1046/j.1365-2133.2002.04669.x. PMID 11966687
- [Background] Di Girolamo N, Chui J, Coroneo MT, Wakefield D. Pathogenesis of pterygia: role of cytokines, growth factors, and matrix metalloproteinases. Prog Retin Eye Res. 2004 Mar;23(2):195-228. doi: 10.1016/j.preteyeres.2004.02.002. PMID 15094131
- [Background] Tan DT, Lim AS, Goh HS, Smith DR. Abnormal expression of the p53 tumor suppressor gene in the conjunctiva of patients with pterygium. Am J Ophthalmol. 1997 Mar;123(3):404-5. doi: 10.1016/s0002-9394(14)70141-2. PMID 9063255
- [Background] Tan DT, Chee SP, Dear KB, Lim AS. Effect of pterygium morphology on pterygium recurrence in a controlled trial comparing conjunctival autografting with bare sclera excision. Arch Ophthalmol. 1997 Oct;115(10):1235-40. doi: 10.1001/archopht.1997.01100160405001. PMID 9338666
- [Background] Prabhasawat P, Barton K, Burkett G, Tseng SC. Comparison of conjunctival autografts, amniotic membrane grafts, and primary closure for pterygium excision. Ophthalmology. 1997 Jun;104(6):974-85. doi: 10.1016/s0161-6420(97)30197-3. PMID 9186439
- [Background] Ang LP, Chua JL, Tan DT. Current concepts and techniques in pterygium treatment. Curr Opin Ophthalmol. 2007 Jul;18(4):308-13. doi: 10.1097/ICU.0b013e3281a7ecbb. PMID 17568207
- [Background] Prabhasawat P, Tesavibul N, Leelapatranura K, Phonjan T. Efficacy of subconjunctival 5-fluorouracil and triamcinolone injection in impending recurrent pterygium. Ophthalmology. 2006 Jul;113(7):1102-9. doi: 10.1016/j.ophtha.2006.02.026. Epub 2006 May 26. PMID 16730066
- [Background] Hirst LW, Sebban A, Chant D. Pterygium recurrence time. Ophthalmology. 1994 Apr;101(4):755-8. doi: 10.1016/s0161-6420(94)31270-x. PMID 8152771
- [Background] Razeghinejad MR, Hosseini H, Ahmadi F, Rahat F, Eghbal H. Preliminary results of subconjunctival bevacizumab in primary pterygium excision. Ophthalmic Res. 2010;43(3):134-8. doi: 10.1159/000252980. Epub 2009 Oct 29. PMID 19887878
- [Background] Poenaru Sava MG, Raica ML, Cimpean AM. VEGF mRNA assessment in human pterygium: a new 'scope' for a future hope. Ophthalmic Res. 2014;52(3):130-5. doi: 10.1159/000363142. Epub 2014 Oct 3. PMID 25300614
- [Background] Mansour AM. Treatment of inflamed pterygia or residual pterygial bed. Br J Ophthalmol. 2009 Jul;93(7):864-5. doi: 10.1136/bjo.2008.155291. PMID 19553512
- [Background] Teng CC, Patel NN, Jacobson L. Effect of subconjunctival bevacizumab on primary pterygium. Cornea. 2009 May;28(4):468-70. doi: 10.1097/ICO.0b013e31818d382d. PMID 19411971
- [Background] Wu PC, Kuo HK, Tai MH, Shin SJ. Topical bevacizumab eyedrops for limbal-conjunctival neovascularization in impending recurrent pterygium. Cornea. 2009 Jan;28(1):103-4. doi: 10.1097/ICO.0b013e3181822615. PMID 19092418
- [Result] Hosseini H, Nejabat M, Khalili MR. Bevacizumab (Avastin) as a potential novel adjunct in the management of pterygia. Med Hypotheses. 2007;69(4):925-7. doi: 10.1016/j.mehy.2007.01.047. Epub 2007 Mar 26. PMID 17367957
- [Result] Hurmeric V, Vaddavalli P, Galor A, Perez VL, Roman JS, Yoo SH. Single and multiple injections of subconjunctival ranibizumab for early, recurrent pterygium. Clin Ophthalmol. 2013;7:467-73. doi: 10.2147/OPTH.S40400. Epub 2013 Mar 4. PMID 23486999
- [Result] Galor A, Yoo SH, Piccoli FV, Schmitt AJ, Chang V, Perez VL. Phase I study of subconjunctival ranibizumab in patients with primary pterygium undergoing pterygium surgery. Am J Ophthalmol. 2010 Jun;149(6):926-931.e2. doi: 10.1016/j.ajo.2010.01.015. Epub 2010 Apr 24. PMID 20417925
- [Result] Mandalos A, Tsakpinis D, Karayannopoulou G, Tsinopoulos I, Karkavelas G, Chalvatzis N, Dimitrakos S. The effect of subconjunctival ranibizumab on primary pterygium: a pilot study. Cornea. 2010 Dec;29(12):1373-9. doi: 10.1097/ICO.0b013e3181d927b9. PMID 20856107
- [Result] Benayoun Y, Adenis JP, Casse G, Forte R, Robert PY. Effects of subconjunctival bevacizumab on corneal neovascularization: results of a prospective study. Cornea. 2012 Aug;31(8):937-44. doi: 10.1097/ICO.0b013e31823f8d71. PMID 22357391
- [Result] Enkvetchakul O, Thanathanee O, Rangsin R, Lekhanont K, Suwan-Apichon O. A randomized controlled trial of intralesional bevacizumab injection on primary pterygium: preliminary results. Cornea. 2011 Nov;30(11):1213-8. doi: 10.1097/ICO.0b013e31821c9b44. PMID 21915047
- [Result] Lekhanont K, Patarakittam T, Thongphiew P, Suwan-apichon O, Hanutsaha P. Randomized controlled trial of subconjunctival bevacizumab injection in impending recurrent pterygium: a pilot study. Cornea. 2012 Feb;31(2):155-61. doi: 10.1097/ICO.0b013e3182151e0e. PMID 22081150
- [Result] Razeghinejad MR, Banifatemi M. Subconjunctival bevacizumab for primary pterygium excision; a randomized clinical trial. J Ophthalmic Vis Res. 2014 Jan;9(1):22-30. PMID 24982728
- [Result] Razeghinejad R, Banifatemi M, Hosseini H. The effect of different doses of subconjunctival bevacizumab on the recurrence rate of excised primary pterygium. Bull Soc Belge Ophtalmol. 2013;(322):13-20. PMID 24923077
- [Result] Shenasi A, Mousavi F, Shoa-Ahari S, Rahimi-Ardabili B, Fouladi RF. Subconjunctival bevacizumab immediately after excision of primary pterygium: the first clinical trial. Cornea. 2011 Nov;30(11):1219-22. doi: 10.1097/ICO.0b013e31820ca63f. PMID 21955635
- [Result] Shahin MM, Elbendary AM, Elwan MM. Intraoperative subconjunctival bevacizumab as an adjunctive treatment in primary pterygium: a preliminary report. Ophthalmic Surg Lasers Imaging. 2012 Nov-Dec;43(6):459-66. doi: 10.3928/15428877-20120802-02. Epub 2012 Aug 10. PMID 22882007
- [Result] Ozgurhan EB, Agca A, Kara N, Yuksel K, Demircan A, Demirok A. Topical application of bevacizumab as an adjunct to recurrent pterygium surgery. Cornea. 2013 Jun;32(6):835-8. doi: 10.1097/ICO.0b013e3182772d4e. PMID 23187164
- [Result] Karalezli A, Kucukerdonmez C, Akova YA, Koktekir BE. Does topical bevacizumab prevent postoperative recurrence after pterygium surgery with conjunctival autografting? Int J Ophthalmol. 2014 Jun 18;7(3):512-6. doi: 10.3980/j.issn.2222-3959.2014.03.23. eCollection 2014. PMID 24967201
- [Result] Nava-Castaneda A, Olvera-Morales O, Ramos-Castellon C, Garnica-Hayashi L, Garfias Y. Randomized, controlled trial of conjunctival autografting combined with subconjunctival bevacizumab for primary pterygium treatment: 1-year follow-up. Clin Exp Ophthalmol. 2014 Apr;42(3):235-41. doi: 10.1111/ceo.12140. Epub 2013 Jul 5. PMID 23777441
- [Result] Hu Q, Qiao Y, Nie X, Cheng X, Ma Y. Bevacizumab in the treatment of pterygium: a meta-analysis. Cornea. 2014 Feb;33(2):154-60. doi: 10.1097/ICO.0000000000000037. PMID 24326333
- [Result] Bahar I, Kaiserman I, McAllum P, Rootman D, Slomovic A. Subconjunctival bevacizumab injection for corneal neovascularization in recurrent pterygium. Curr Eye Res. 2008 Jan;33(1):23-8. doi: 10.1080/02713680701799101. PMID 18214740
- [Result] Bayar SA, Kucukerdonmez C, Oner O, Akova YA. Subconjunctival bevacizumab in the impending recurrent pterygia. Int Ophthalmol. 2014 Jun;34(3):541-7. doi: 10.1007/s10792-013-9852-1. Epub 2013 Sep 12. PMID 24026871
- [Result] Fallah Tafti MR, Khosravifard K, Mohammadpour M, Hashemian MN, Kiarudi MY. Efficacy of intralesional bevacizumab injection in decreasing pterygium size. Cornea. 2011 Feb;30(2):127-9. doi: 10.1097/ICO.0b013e3181e16d67. PMID 20885313
- [Result] Besharati MR, Manaviat MR, Souzani A. Subconjunctival bevacizumab injection in treatment of pterygium. Acta Med Iran. 2011;49(3):179-83. PMID 21681707
- [Result] Sarac O, Demirel S, Oltulu R. Efficacy of intralesional bevacizumab administration in primary pterygium: a quantitative analysis. Eye Contact Lens. 2014 Jan;40(1):46-50. doi: 10.1097/ICL.0000000000000004. PMID 24335454
- [Result] Kocabora SM, Fazil K, Ozsutcu M, Doyduk-Kocabora A, Gulkilik G. Subconjunctival bevacizumab injection in the surgery of primary pterygium: comparison with intraoperative mitomycin-C. Bull Soc Belge Ophtalmol. 2013;(322):7-12. PMID 24923076